CLINICAL TRIAL: NCT02384356
Title: A Longitudinal Survey of Health in Bolivia
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist, Professor of Health Behavior and Health Education and of Internal Medicine, University of Michigan
Other Study IDs: HUM00071766
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Chronic Disease
Keywords: Non-communicable diseases; Chronic disease; Mobile health; Diabetes Mellitus; Hypertension; Bolivia; Longitudinal survey; Health indicators; Primary care; Ambulatory care
MeSH Terms: conditions — Chronic Disease; Noncommunicable Diseases; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to gather baseline surveillance data about the current health status of adults with chronic health conditions in La Paz and El Alto, Bolivia and identify barriers to the management of NCDs during face-to-face outpatient encounters as well as via novel mobile health services.

DETAILED DESCRIPTION:
Within Latin America, there is a significant lack of data about the medical management and self-care for patients with non-communicable diseases (NCDs), such as diabetes and hypertension. In an effort to improve availability of such data in the Latin American region, the World Health Organization (WHO) created and tailored a survey tool that has been used in various countries throughout Central and South America. Our own research team has extensive experience surveying clinic-based populations in Latin America regarding their chronic disease burden and the potential effectiveness of novel approaches to self-care support via mobile phones. The objective of the planned project is to gather baseline surveillance data for non-communicable diseases in urban and peri-urban Bolivian communities, using the WHO instrument as a foundation with modifications to reflect local public health priorities and the goal of developing mobile health services that improve self-management support.

This project will be conducted by investigators and students of the University of Michigan Schools of Medicine, Public Health, and Information, in partnership with the Catholic University of Bolivia, San Pablo (UCB-San Pablo). The over-arching aim is to conduct a longitudinal survey of health indicators in a variety of primary and ambulatory care sites within clinics associated with Universidad Católica Boliviana, including SEDES La Paz and Universidad Mayor San Andres, in La Paz and El Alto, Bolivia. The survey is based on: a) the World Health Organizations' Division of Disease Prevention and Control's Program on Non-Communicable Diseases' (NCD) Surveillance Toolkit: Risk Factors for Non-Communicable Diseases, with the addition of b) the 8 Item Patient Health Questionnaire (PHQ-8) to screen for Depression, c) the Alcohol Use Disorders Identification Test (AUDIT), d) the Patient Assessment of Chronic Illness Care (PACIC) Questionnaire, e) questions developed by our research team regarding the feasibility and desirability of mobile health monitoring and self-care support and f) 8 item Morisky Medication use questions. By using validated survey instruments, the investigators will be able to compare health indicators across countries and provide the participating Bolivian government agencies and universities information crucial to understanding the factors contributing to the development and maintenance of NCD services in Bolivia. Specifically, this study will provide baseline data, which does not exist to date, identifying the prevalent risk factors for NCDs and the barriers to those patients' care. More generally, the investigators will gain invaluable experience regarding the feasibility of enrolling large representative samples in various outpatient sites for use in subsequent observational studies of NCD management and in randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Existing diagnosis (per medical record) of at least 1 chronic health issue: diabetes, hypertension, cardiac issues, angina, high cholesterol, depression, cancer, stroke, arthritis, chronic bronchitis, emphysema, COPD, migraine headaches, heartburn, acid reflux or irritable bowel syndrome, stomach or duodenal ulcers, chronic back pain or sciatica, asthma, history of gestational diabetes (female), history of polycystic ovary syndrome (female)
* If no existing diagnosis of at least 1 chronic health issue, then clinical indicator patient may be at risk of diabetes (has a close relative with diabetes, female patient who delivered a baby weighing more than 9 pounds); PHQ-2 score between 3-6, BMI >25; or, Systolic BP over 140

Exclusion Criteria:

* Life-threatening health problem such as cancer with less than a six month life expectancy
* Are visiting the clinic for an urgent health problem (for themselves)
* If they have severe mental illness as reported by their clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients visiting clinics associated with Universidad Católica Boliviana, including SEDES La Paz and Universidad Mayor San Andres, in La Paz and El Alto, Bolivia for a non-urgent health problem.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Health Status using general health-related quality of life, perceived health, and PHQ8 | Baseline and then annually for up to 7 years
  Outcomes will be assessed at baseline and follow-up if follow-up is possible.

SECONDARY OUTCOMES:
Demographics, use of formal care and access, substance use, NCD diagnoses, self-care behavior, knowledge/perceptions, and anthropometric measures | Baseline and then annually for up to 7 years
  Information will be gathered at baseline and follow-up to assess changes in status.

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (2):
- Bolivia (2):
  - Universidad Católica Boliviana associated clinics, including SEDES La Paz and Universidad Mayor San Andres, El Alto
  - Universidad Católica Boliviana associated clinics, including SEDES La Paz and Universidad Mayor San Andres, La Paz

IPD SHARING:
Plan to Share IPD: No